CLINICAL TRIAL: NCT05029167
Title: REstrictive Versus LIberal Oxygen Strategy and Its Effect on Pulmonary Hypertension After Out-of-hospital Cardiac Arrest (RELIEPH-study): a Substudy Protocol for a Randomised Clinical Trial
Brief Title: REstrictive Versus LIberal Oxygen Strategy and Its Effect on Pulmonary Hypertension After Out-of-hospital Cardiac Arrest (RELIEPH-study)
Acronym: RELIEPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-2021xxxx
Record Dates: First submitted 2021-08-11; First posted 2021-08-31 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hypertension, Pulmonary Arterial; Out-Of-Hospital Cardiac Arrest; Intensive Care Unit; Oxygen Therapy; Mechanical Ventilation; Resuscitation
Keywords: Out-of-hospital cardiac arrest; Resuscitation; Oxygen; Intensive Care Unit; Mechanical ventilation; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Out-of-Hospital Cardiac Arrest; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: The RELIEPH trial is a substudy of the BOX trial, which is a multicenter, randomised clinical trial with a 2x2 factorial design. Patients are allocated 1:1:1:1 to two interventions, respectively high- or low mean arterial pressures (double blinded) and restrictive- or liberal oxygenation (open label). The RELIEPH trial focuses on the oxygen intervention and only has access to data from one trial site. This makes the RELIEPH trial a single-center, parallel-group randomised controlled trial with patients allocated 1:1 to the oxygen target interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Restrictive PaO2 and low normal MAP (Active Comparator): Patients receiving PaO2 9-10 kPa (68-75 mmHg) and MAP 63 mmHg during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: Restrictive PaO2; Other: Low normal MAP
- Restrictive PaO2 and high normal MAP (Active Comparator): Patients receiving PaO2 9-10 kPa (68-75 mmHg) and MAP 77 mmHg during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: Restrictive PaO2; Other: High normal MAP
- Liberal PaO2 and low normal MAP (Active Comparator): Patients receiving PaO2 13-14 kPa (98-105 mmHg) and MAP 63 mmHg during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: Low normal MAP; Other: Liberal PaO2
- Liberal PaO2 and high normal MAP (Active Comparator): Patients receiving PaO2 13-14 kPa (98-105 mmHg) and MAP 77 mmHg during targeted temperature management (36 hours) after OHCA.
  Interventions: Other: Liberal PaO2; Other: High normal MAP

INTERVENTIONS:
Other: Restrictive PaO2 — Patients are randomized to a PaO2 target of 9-10 kPa (open-label).
  Other Names: PaO2 target at 9-10 kPa.
  Arms: Restrictive PaO2 and high normal MAP; Restrictive PaO2 and low normal MAP
Other: Low normal MAP — The patients are randomized to receive a Phillips M1006B blood pressure measuring module, offset by +10 %. All patients will target a MAP of 70, but due to the offset module, the patients will target an actual blood pressure of 63 mmHg.
  Other Names: Mean arterial blood pressure at 63 mmHg.
  Arms: Liberal PaO2 and low normal MAP; Restrictive PaO2 and low normal MAP
Other: Liberal PaO2 — Patients are randomized to a PaO2 target of 13-14 kPa (open-label).
  Other Names: PaO2 target at 13-14 kPa.
  Arms: Liberal PaO2 and high normal MAP; Liberal PaO2 and low normal MAP
Other: High normal MAP — The patients are randomized to receive a Phillips M1006B blood pressure measuring module, offset by -10 %. All patients will target a MAP of 70, but due to the offset module, the patients will target an actual blood pressure of 77mmHg.
  Other Names: Mean arterial blood pressure at 77 mmHg.
  Arms: Liberal PaO2 and high normal MAP; Restrictive PaO2 and high normal MAP

SUMMARY:
Background: For patients with out-of-hospital cardiac arrest (OHCA) at the intensive care unit (ICU), oxygen therapy plays an important role in post resuscitation care. During hospitalisation, a lot of these patients occur with pulmonary arterial hypertension (PAH). Currently a wide oxygen target is recommended but no evidence regarding optimal treatment targets to minimise the prevalence of PAH exists.

Methods: The RELIEPH trial is a substudy within the BOX (Blood pressure and OXygenation targets in post resuscitation care) trial. It is a single-center, parallel-group randomised controlled clinical trial. 300 patients with OHCA hospitalised at the ICU are allocated to one of the two oxygenation interventions, either a restrictive- (9-10 kPa) or liberal (13-14 kPa) oxygen target both within the recommended range. The primary outcome is the fraction of time with pulmonary hypertension (mPAP >25 mmHg) out of total time with mechanical ventilation. Secondary outcomes are: length of ICU stay among survivors, lactate clearance, right ventricular failure, 30 days mortality and plasma brain natriuretic peptide (BNP) level 48 hours from randomisation.

Discussion: This study hypothesises that a liberal target of oxygen reduces the time with PAH during mechanical ventilation compared to a restrictive oxygen target in patients with OHCA at the ICU. When completed, this study hopes to provide new knowledge regarding which oxygen target is beneficial for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* OHCA of presumed cardiac cause
* Sustained ROSC
* Unconsciousness (Glasgow coma scale <8) after sustained ROSC

Exclusion Criteria:

* Conscious patients (obeying verbal commands)
* Females of childbearing potential (unless a negative HCG test can rule out pregnancy within the inclusion window)
* In-hospital cardiac arrest
* OHCA of presumed non-cardiac cause e.g. after trauma or dissection/rupture of major artery or cardiac arrest caused by initial hypoxia (i.e. drowning, suffocation, hanging).
* Known bleeding diathesis (medically induced coagulopathy (e.g. warfarin, NOAC, clopidogrel) does not exclude the patient)
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed acute stroke
* Unwitnessed asystole
* Known limitations in therapy and Do Not Resuscitate-order
* Known disease making 180 days survival unlikely
* Known pre-arrest cerebral performance category 3 or 4
* >4 hours (240 minutes) from ROSC to screening
* Systolic blood pressure <80 mmHg in spite of fluid loading/vasopressor and/or inotropic medication/intra-aortic balloon pump/axial flow device
* Temperature on admission <30°C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary hypertension | Up to 30 days.
  Fraction of time with pulmonary hypertension (mPAP >25 mmHg) out of total time with mechanical ventilation.

SECONDARY OUTCOMES:
Length of ICU stay. | Up to 8 weeks.
  Length of ICU stay among survivors.
Lactate clearance. | 24 hours.
  >30% reduction in lactate level.
Right ventricular failure. | Up to 8 weeks.
  Cardiac index <2 and central venous pressure >18 mmHg.
Mortality. | 30 days after ROSC.
  Dead or alive.
Plasma brain natriuretic peptide. | 48 hours from randomisation.
  Plasma brain natriuretic peptide level.

CONTACTS AND LOCATIONS:
Locations (1):
- Depart med Cardiothoracic Intensive Care, Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in post-resuscitation care. Data or samples shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement.

REFERENCES:
- [Background] Zhang Z, Xu X. Lactate clearance is a useful biomarker for the prediction of all-cause mortality in critically ill patients: a systematic review and meta-analysis*. Crit Care Med. 2014 Sep;42(9):2118-25. doi: 10.1097/CCM.0000000000000405. PMID 24797375
- [Background] Young P, Bailey M, Bellomo R, Bernard S, Dicker B, Freebairn R, Henderson S, Mackle D, McArthur C, McGuinness S, Smith T, Swain A, Weatherall M, Beasley R. HyperOxic Therapy OR NormOxic Therapy after out-of-hospital cardiac arrest (HOT OR NOT): a randomised controlled feasibility trial. Resuscitation. 2014 Dec;85(12):1686-91. doi: 10.1016/j.resuscitation.2014.09.011. Epub 2014 Sep 28. PMID 25261605
- [Background] Yamamoto R, Yoshizawa J. Oxygen administration in patients recovering from cardiac arrest: a narrative review. J Intensive Care. 2020 Aug 12;8:60. doi: 10.1186/s40560-020-00477-w. eCollection 2020. PMID 32832091
- [Background] Simonneau G, Gatzoulis MA, Adatia I, Celermajer D, Denton C, Ghofrani A, Gomez Sanchez MA, Krishna Kumar R, Landzberg M, Machado RF, Olschewski H, Robbins IM, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D34-41. doi: 10.1016/j.jacc.2013.10.029. PMID 24355639
- [Background] Schjorring OL, Klitgaard TL, Perner A, Wetterslev J, Lange T, Siegemund M, Backlund M, Keus F, Laake JH, Morgan M, Thormar KM, Rosborg SA, Bisgaard J, Erntgaard AES, Lynnerup AH, Pedersen RL, Crescioli E, Gielstrup TC, Behzadi MT, Poulsen LM, Estrup S, Laigaard JP, Andersen C, Mortensen CB, Brand BA, White J, Jarnvig IL, Moller MH, Quist L, Bestle MH, Schonemann-Lund M, Kamper MK, Hindborg M, Hollinger A, Gebhard CE, Zellweger N, Meyhoff CS, Hjort M, Bech LK, Grofte T, Bundgaard H, Ostergaard LHM, Thyo MA, Hildebrandt T, Uslu B, Solling CG, Moller-Nielsen N, Brochner AC, Borup M, Okkonen M, Dieperink W, Pedersen UG, Andreasen AS, Buus L, Aslam TN, Winding RR, Schefold JC, Thorup SB, Iversen SA, Engstrom J, Kjaer MN, Rasmussen BS; HOT-ICU Investigators. Lower or Higher Oxygenation Targets for Acute Hypoxemic Respiratory Failure. N Engl J Med. 2021 Apr 8;384(14):1301-1311. doi: 10.1056/NEJMoa2032510. Epub 2021 Jan 20. PMID 33471452
- [Background] Panwar R, Hardie M, Bellomo R, Barrot L, Eastwood GM, Young PJ, Capellier G, Harrigan PW, Bailey M; CLOSE Study Investigators; ANZICS Clinical Trials Group. Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Jan 1;193(1):43-51. doi: 10.1164/rccm.201505-1019OC. PMID 26334785
- [Background] Nolan JP, Soar J, Cariou A, Cronberg T, Moulaert VR, Deakin CD, Bottiger BW, Friberg H, Sunde K, Sandroni C; European Resuscitation Council; European Society of Intensive Care Medicine. European Resuscitation Council and European Society of Intensive Care Medicine 2015 guidelines for post-resuscitation care. Intensive Care Med. 2015 Dec;41(12):2039-56. doi: 10.1007/s00134-015-4051-3. PMID 26464394
- [Background] Nash G, Blennerhassett JB, Pontoppidan H. Pulmonary lesions associated with oxygen therapy and artificial ventilation. N Engl J Med. 1967 Feb 16;276(7):368-74. doi: 10.1056/NEJM196702162760702. No abstract available. PMID 6017244
- [Background] Moudgil R, Michelakis ED, Archer SL. Hypoxic pulmonary vasoconstriction. J Appl Physiol (1985). 2005 Jan;98(1):390-403. doi: 10.1152/japplphysiol.00733.2004. PMID 15591309
- [Background] McLaughlin VV, Shah SJ, Souza R, Humbert M. Management of pulmonary arterial hypertension. J Am Coll Cardiol. 2015 May 12;65(18):1976-97. doi: 10.1016/j.jacc.2015.03.540. PMID 25953750
- [Background] Luecke T, Pelosi P. Clinical review: Positive end-expiratory pressure and cardiac output. Crit Care. 2005;9(6):607-21. doi: 10.1186/cc3877. Epub 2005 Oct 18. PMID 16356246
- [Background] Kirkegaard H, Taccone FS, Skrifvars M, Soreide E. Postresuscitation Care after Out-of-hospital Cardiac Arrest: Clinical Update and Focus on Targeted Temperature Management. Anesthesiology. 2019 Jul;131(1):186-208. doi: 10.1097/ALN.0000000000002700. PMID 31021845
- [Background] Huynh TN, Weigt SS, Sugar CA, Shapiro S, Kleerup EC. Prognostic factors and outcomes of patients with pulmonary hypertension admitted to the intensive care unit. J Crit Care. 2012 Dec;27(6):739.e7-13. doi: 10.1016/j.jcrc.2012.08.006. Epub 2012 Oct 22. PMID 23089677
- [Background] Grasner JT, Lefering R, Koster RW, Masterson S, Bottiger BW, Herlitz J, Wnent J, Tjelmeland IB, Ortiz FR, Maurer H, Baubin M, Mols P, Hadzibegovic I, Ioannides M, Skulec R, Wissenberg M, Salo A, Hubert H, Nikolaou NI, Loczi G, Svavarsdottir H, Semeraro F, Wright PJ, Clarens C, Pijls R, Cebula G, Correia VG, Cimpoesu D, Raffay V, Trenkler S, Markota A, Stromsoe A, Burkart R, Perkins GD, Bossaert LL; EuReCa ONE Collaborators. EuReCa ONE-27 Nations, ONE Europe, ONE Registry: A prospective one month analysis of out-of-hospital cardiac arrest outcomes in 27 countries in Europe. Resuscitation. 2016 Aug;105:188-95. doi: 10.1016/j.resuscitation.2016.06.004. Epub 2016 Jun 16. PMID 27321577
- [Background] Gomersall CD, Joynt GM, Freebairn RC, Lai CK, Oh TE. Oxygen therapy for hypercapnic patients with chronic obstructive pulmonary disease and acute respiratory failure: a randomized, controlled pilot study. Crit Care Med. 2002 Jan;30(1):113-6. doi: 10.1097/00003246-200201000-00018. PMID 11905405
- [Background] Girardis M, Busani S, Damiani E, Donati A, Rinaldi L, Marudi A, Morelli A, Antonelli M, Singer M. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1583-1589. doi: 10.1001/jama.2016.11993. PMID 27706466
- [Background] de Jonge E, Peelen L, Keijzers PJ, Joore H, de Lange D, van der Voort PH, Bosman RJ, de Waal RA, Wesselink R, de Keizer NF. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care. 2008;12(6):R156. doi: 10.1186/cc7150. Epub 2008 Dec 10. PMID 19077208
- [Background] Asfar P, Schortgen F, Boisrame-Helms J, Charpentier J, Guerot E, Megarbane B, Grimaldi D, Grelon F, Anguel N, Lasocki S, Henry-Lagarrigue M, Gonzalez F, Legay F, Guitton C, Schenck M, Doise JM, Devaquet J, Van Der Linden T, Chatellier D, Rigaud JP, Dellamonica J, Tamion F, Meziani F, Mercat A, Dreyfuss D, Seegers V, Radermacher P; HYPER2S Investigators; REVA research network. Hyperoxia and hypertonic saline in patients with septic shock (HYPERS2S): a two-by-two factorial, multicentre, randomised, clinical trial. Lancet Respir Med. 2017 Mar;5(3):180-190. doi: 10.1016/S2213-2600(17)30046-2. Epub 2017 Feb 15. PMID 28219612
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- See also: Blood Pressure and OXygenation Targets After OHCA — http://clinicaltrials.gov/show/NCT03141099